CLINICAL TRIAL: NCT00906425
Title: Randomized, Controlled Clinical Study Comparing Submerged vs. Trans-mucosal Placement of P.004 Implants in the Anterior Maxilla and Mandible by Evaluation of the Change in Bone Level Between 1st Stage Surgery and 6 Months Post Surgery
Brief Title: Clinical Study Comparing Submerged Versus Trans-mucosal Healing of P.004 Implants in the Anterior Mandible and Maxilla
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR 05/05
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Jaw, Edentulous, Partially
Keywords: Dental Implant
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Submerged healing (Active Comparator): The Straumann Bone Level Implant(s) will be placed using a submerged healing treatment
  Interventions: Device: Straumann Bone Level Implant
- Trans-mucosal healing (Active Comparator): The Straumann Bone Level Implant(s) will be placed using a trans-mucosal healing treatment
  Interventions: Device: Straumann Bone Level Implant

INTERVENTIONS:
Device: Straumann Bone Level Implant — Straumann Bone Level Implant, SLActive surface, diameter 4.1, length 8, 10, 12, and 14 mm

SUMMARY:
The purpose of this study is To demonstrate that there is no difference in change in bone level around P.004 implants between 1st stage surgery and 6 months post surgery when transmucosal implant placement is compared to submerged implant placement

DETAILED DESCRIPTION:
The primary objective of this study is to determine the level at which the bone can be maintained in relation to the implant shoulder for the P.004 two-stage implant when placed in a submerged or a trans-mucosal procedure in single tooth gaps in the anterior region. The primary parameter will be measured by radiography 26 weeks after loading of the implant.

ELIGIBILITY:
Inclusion Criteria:

* Males and females >18 years of age.
* Implant placement planned in the anterior maxilla or mandible (FDI tooth numbers 21 - 25, 11 - 15, 31-35, 41-45).
* Tooth site must have a natural tooth both mesially and distally in the adjacent tooth positions
* Opposing dentition of natural teeth, or tooth or implant-supported fixed restorations.
* Adequate bone quality and quantity at the implant site to permit the insertion of a Straumann P.004 SLActive implant of 8, 10, 12, or 14 mm length.
* Presence of a sufficient band of keratinized mucosa (min. 2 mm) to allow surgical manipulation and suturing according to the protocol
* Signed informed consent document before being treated in the study

Exclusion Criteria:

* Systemic disease that would interfere with dental implant therapy (e.g. uncontrolled diabetes)
* Any contraindications for oral surgical procedures
* Current untreated periodontitis or gingivitis
* Probing pocket depth of more than 4 mm at one of the adjacent teeth
* Mucosal diseases (e.g. erosive lichen planus)
* History of local irradiation therapy
* Bone augmentation procedures if the procedure require healing time of more than 12 weeks after implant placement
* Implants in adjacent position to planned implant
* Severe bruxing or clenching habits
* Heavy smokers: Patients who smoke more than 20 cigarettes per day
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation.
* Patients with inadequate oral hygiene or unmotivated for adequate home care

Secondary Exclusion Criteria at Implant Surgery:

* Lack of primary stability of the implant
* Inappropriate implant position to insert implants according to the prosthetic requirements.
* Patients with augmentation procedures requiring more than 12 weeks healing time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2006-10; Primary Completion 2008-06 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hammerle, Principal Investigator — University of Zurich
Locations (11):
- United States (2):
  - Dr. Jeffery Ganeles, Boca Raton, Florida
  - Dr. William C. Martin, Gainesville, Florida
- Dr. Stephen T. Chen, Melbourne, Australia
- Germany (4):
  - Prof. Wiltfang, Kiel, Schleswig-Holstein
  - Michael Gahlert, München
  - Katharinenhospital, Stuttgart
  - Private Universität Witten/ Herdecke, Witten/ Herdecke
- Dr. Luca Cordaro, Rome, Italy
- Prof. Mariano Sanz, Madrid, Spain
- Dr. Carl-Johan Ivanoff, Mölndal, Sweden
- Christoph Hämmerle, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hammerle CHF, Jung RE, Sanz M, Chen S, Martin WC, Jackowski J; this multicenter study group; Ivanoff CJ, Cordaro L, Ganeles J, Weingart D, Wiltfang J, Gahlert M. Submerged and transmucosal healing yield the same clinical outcomes with two-piece implants in the anterior maxilla and mandible: interim 1-year results of a randomized, controlled clinical trial. Clin Oral Implants Res. 2012 Feb;23(2):211-219. doi: 10.1111/j.1600-0501.2011.02210.x. Epub 2011 Jul 4. PMID 21722188
- [Result] Cordaro L, Torsello F, Chen S, Ganeles J, Bragger U, Hammerle C. Implant-supported single tooth restoration in the aesthetic zone: transmucosal and submerged healing provide similar outcome when simultaneous bone augmentation is needed. Clin Oral Implants Res. 2013 Oct;24(10):1130-6. doi: 10.1111/j.1600-0501.2012.02521.x. Epub 2012 Jun 15. PMID 22697581

RESULTS

PARTICIPANT FLOW:
Groups:
- Submerged Healing: The dental implants will be placed using a submerged healing treatment
- Trans-mucosal Healing: The dental implants will be placed using a trans-mucosal healing treatment
Period: Overall Study
Arm/Group | Submerged Healing | Trans-mucosal Healing
Started | 73 | 72
6 Months | 69 (ITT population) | 64 (ITT population)
1 Year | 67 (ITT population) | 60 (ITT population)
2 Year | 62 (ITT population) | 58 (ITT population)
Completed | 0 (Clinical Trial expected to be completed in 2013) | 0 (Clinical Trial expected to be completed in 2013)
Not Completed | 73 | 72

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Submerged Healing | Trans-mucosal Healing | Total
Number analyzed (Participants) | 73 | 72 | 145
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 62 | 59 | 121
  >=65 years | 11 | 13 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 31 | 70
  Male | 34 | 41 | 75
Region of Enrollment [Number; unit: participants]
  United States | 14 | 19 | 33
  Spain | 12 | 12 | 24
  Australia | 10 | 9 | 19
  Germany | 18 | 14 | 32
  Switzerland | 7 | 7 | 14
  Italy | 6 | 6 | 12
  Sweden | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Bone Level (Distance B) After 6 Months Compared to Baseline (=Surgery)
Description: The primary aim is to measure the bone level change between mesial and distal aspects of the implant at 6 months post implantation. The reference point for the bone level measurement is the implant shoulder.
Time Frame: Baseline and 6 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Submerged Healing | Trans-mucosal Healing
Number analyzed (Participants) | 65 | 59
millimeters | -0.32 (0.47) | -0.29 (0.35)

2. Secondary Outcome: Implant Survival Rate
Description: The percentage of implants that remain in place in the jaw.
Time Frame: 6 months
Measure: Number; unit: % of implants
Arm/Group | Submerged Healing | Trans-mucosal Healing
Number analyzed (Participants) | 67 | 60
% of implants | 100 | 98.3

3. Secondary Outcome: Implant Survival Rate
Description: The percentage of implants that remain in place in the jaw.
Time Frame: 12 months
Measure: Number; unit: % of implants
Arm/Group | Submerged Healing | Trans-mucosal Healing
Number analyzed (Participants) | 67 | 60
% of implants | 100 | 98.3

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Submerged Healing | Trans-mucosal Healing
Serious Adverse Events (participants affected / at risk) | 2/73 | 0/72
Other Adverse Events (participants affected / at risk) | 8/73 | 10/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Submerged Healing (N=73) | Trans-mucosal Healing (N=72)
Uterine Cancer (Reproductive system and breast disorders) | 1 (1) | 0 (0)
(General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Submerged Healing (N=73) | Trans-mucosal Healing (N=72)
Implant or site related complications (General disorders) | 1 (1) | 0 (0)
Implant mobility (General disorders) | 0 (0) | 1 (1)
Dehiscence at implant site (General disorders) | 0 (0) | 1 (1)
Gingival/Mucosal Problems (General disorders) | 1 (1) | 0 (0)
Fistula (General disorders) | 1 (1) | 1 (1)
Prosthetic Related Complications (General disorders) | 1 (1) | 2 (2)
Lost/Failure (fracture) of an Abutment (General disorders) | 0 (0) | 1 (1)
Loosening of Occlusal Screw (General disorders) | 0 (0) | 1 (1)
Aesthetic Problems (General disorders) | 0 (0) | 1 (1)
Failure of Prosthetic Part (framework) (General disorders) | 1 (1) | 0 (0)
Acrylic or Porcelain Fractures (General disorders) | 0 (0) | 2 (2)
Uterine Cancer (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Local discomfort/pain around the implant site (General disorders) | 0 (0) | 1 (1)
Allergic reaction (General disorders) | 1 (1) | 0 (0)
Membrane Exposure (General disorders) | 0 (0) | 2 (2)
Hyperthyreosis (Endocrine disorders) | 1 (1) | 0 (0)
(General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less